CLINICAL TRIAL: NCT03735771
Title: Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor: A Sequential Allocation Trial to Determine the Optimum Interval Time Between Boluses of a Fixed Volume of 2.5ml of Bupivacaine 0.25% Plus Fentanyl 8 mcg/ml
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-08
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Labor Pain
Keywords: Epidural; Labor analgesia; Programmed intermittent epidural bolus
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 60 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 60-minute interval. The bolus will consist of 2.5mL of 0.25% Bupivacaine plus fentanyl 8mcg/ml. A PCEA bolus of 2.5mL of 0.25% Bupivacaine plus fentanyl 8mcg/ml will also be available.
  Interventions: Drug: Bupivacaine
- 50 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 50-minute interval. The bolus will consist of 2.5mL of 0.25% Bupivacaine plus fentanyl 8mcg/ml. A PCEA bolus of 2.5mL of 0.25% Bupivacaine plus fentanyl 8mcg/ml will also be available.
  Interventions: Drug: Bupivacaine
- 40 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 40-minute interval. The bolus will consist of 2.5mL of 0.25% Bupivacaine plus fentanyl 8mcg/ml. A PCEA bolus of 2.5mL of 0.25% Bupivacaine plus fentanyl 8mcg/ml will also be available.
  Interventions: Drug: Bupivacaine
- 30 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 30-minute interval. The bolus will consist of 2.5mL of 0.25% Bupivacaine plus fentanyl 8mcg/ml. A PCEA bolus of 2.5mL of 0.25% Bupivacaine plus fentanyl 8mcg/ml will also be available.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 0.25% bupivacaine plus fentanyl 8 mcg/ml
  Other Names: Marcaine

SUMMARY:
Programmed intermittent epidural bolus (PIEB) is a technique of epidural analgesia in which boluses of local anesthetic solutions are injected into the epidural space at a fixed time interval. Despite the increasingly popular use of PIEB for labor analgesia, the optimum regimen of drug delivery has yet to be determined. The outcomes of a chosen regimen will depend on the local anesthetic solution used (drug, concentration and mass) and the parameters established for the PIEB, typically associated with patient controlled epidural analgesia (PCEA). Also, the optimum regimen will depend on the anesthetic and obstetric outcomes of interest.

The investigators have conducted several studies aiming at establishing the optimum PIEB regimen for the patient population at Mount Sinai Hospital. High sensory block levels obtained in some of the previous studies conducted at Mount Sinai Hospital and in other studies in the literature, in spite of not determining adverse effects, suggest an imperfect use of the technique, with an exaggerated and unnecessary spread of the epidural mixture. It is possible that by limiting the spread of the local anesthetic mixture, better analgesia can be provided with less overall consumption of local anesthetic. The investigators wanted to conduct a study using boluses of 2.5 mL of bupivacaine 0.25% with fentanyl 8 mcg/mL. This would maintain the same dose of local anesthetic used in previous studies, but in a much smaller volume. This concentration and volume of bupivacaine has not been tried before as a PIEB regimen.

The hypothesis of this study is that the optimum interval time between PIEB boluses of 2.5 mL of 0.25% bupivacaine plus fentanyl 8 mcg/ml will be between 30 and 60 minutes.

DETAILED DESCRIPTION:
The investigators have conducted several studies aimed at establishing the optimum PIEB regimen for the patient population at Mount Sinai Hospital. The first study was to determine the effective interval of PIEB in 90% of women during first stage of labor (EI90), while using a fixed bolus of 10 mL of bupivacaine 0.0625% with fentanyl 2 μg/mL. This study showed that the PIEB time interval to provide effective analgesia is approximately 40 minutes, which corresponds to an hourly consumption of 9.4 mg of bupivacaine. In that study, however, 44% of the women experienced sensory blocks to ice above the T6 level (although not associated with motor block or hypotension).

The investigators subsequently conducted another study with the same anesthetic solution and the same PIEB interval of 40 minutes, to determine the effective volume (dose) of local anesthetic to produce the same outcome of effective analgesia without breakthrough pain. The conclusion was that the volume (dose) could not be reduced without compromising efficacy of the technique, and not surprisingly, the sensory block distribution was very similar to that in the first study. The investigators believe that the high sensory block levels obtained the previous studies and in other studies in the literature suggest an imperfect use of the technique, with an exaggerated and unnecessary spread of the epidural mixture. The investigators then conducted a third study to determine the effective time interval between boluses of more concentrated bupivacaine 0.125% 5ml plus fentanyl 2 mcg/ml. The EI90 for boluses of 5ml of bupivacaine 0.125% with fentanyl 2 mcg/mL was found to be approximately 35 minutes. Similar to the two previous studies, the incidence of women exhibiting sensory block to ice >T6 was still high, approximately 58.4%.

This study will further pursue the effect of volume reduction while maintaining the dose of local anesthetic. It may be true that a bolus of 5mL was still too large of a volume to limit the epidural spread. A more limited spread could lead to better usage of the local anesthetic, even reducing its hourly consumption.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status II or III
* Full term (greater than or equal to 37 weeks gestation)
* Nulliparous
* Singleton pregnancy, vertex presentation
* Active labor defined as regular painful contractions occurring at 3-5 minutes and with progressive cervical ripening
* Verbal Numerical Pain Score (VNPS) greater than 5 at requesting epidural analgesia (VNPS 0-10)
* Cervical dilatation between 2 and 5 cm

Exclusion Criteria:

* Any contraindication to epidural anesthesia
* Accidental dural puncture
* Allergy or hypersensitivity to bupivacaine or fentanyl
* Use of pharmacological analgesics within the last 4 hours
* Patient refusal to participate in the trial

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Adequate response of the patient, defined as no request for supplemental analgesia | 6 hours
  Adequate response of the patient, defined as no request for supplemental analgesia (PCEA bolus or clinician administered bolus) until the completion of the first stage of labor or until 6 hours following initiation of the programmed intermittent epidural bolus (PIEB).

SECONDARY OUTCOMES:
Sensory block level | 6 hours
  Sensory block to ice will be assessed bilaterally at the mid-clavicular lines, and the level of block will be one level below that where the patient feels as cold as compared to frontal part of the head or cheek

OTHER OUTCOMES:
Motor block level assessed using Bromage score | 6 hours
  Motor block will be assessed with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle.
Pain score | 6 hours
  Pain score measured hourly using VNRS (0-10)
Hypotension | 6 hours
  A decrease in systolic blood pressure greater than 20% from baseline (defined as an average of 3 readings prior to epidural).

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shatalin D, Arzola C, Downey K, Ye XY, Carvalho JCA. Programmed intermittent epidural bolus for labour analgesia during first stage of labour: a sequential allocation trial to determine the effective interval time between boluses of a fixed volume of 2.5 mL of bupivacaine 0.25% plus fentanyl 8 microg.mL-1. Can J Anaesth. 2021 May;68(5):653-660. doi: 10.1007/s12630-021-01922-6. Epub 2021 Feb 2. PMID 33532993